CLINICAL TRIAL: NCT04403984
Title: Investigation of the Prognostic Value of Genomic Alterations or Protein Expression in Patients With Operated Early Breast Cancer of Luminal A or Luminal B Subtypes
Brief Title: Investigation of Genomic Alteration in Patients With Luminal A or Luminal B Subtypes
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hellenic Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Other Study IDs: HE10A13
Record Dates: First submitted 2020-05-21; First posted 2020-05-27 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer
Keywords: Early breast cancer; Luminal A breast cancer; Luminal B breast cancer; Operated breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Luminal A breast cancer: Patients confirmed with Luminal A breast cancer sub type
- Patients with Luminal B breast cancer: Patients confirmed with Luminal B breast cancer sub type

SUMMARY:
This is a translational study in patients with operated early breast cancer of Luminal A or Luminal B sub types.The Hellenic Cooperative Oncology Group (HeCOG) has designed an observational biomarker-driven study in patients with Luminal A or Luminal B breast cancer, with the aim to collect valuable biological material from these patients and investigate biomarkers with potential prognostic value.

DETAILED DESCRIPTION:
The HE10A/13 study is an observational study of the Hellenic Cooperative Oncology Group (HeCOG). Its main purpose is the collection of biological material from patients in search of prognostic / predictive biomarkers. Each patient signed an informed consent for the provision of biologic material for future research purposes. The study was conducted in accordance with the Declaration of Helsinki. The clinical and translational protocol has been approved by the Hellenic Cooperative Oncology Group Scientific Committee and is under review by the Institutional Review Board of Metropolitan Hospital. Patients exclusively with Luminal A or Luminal B (Estrogen Receptors (ER)-positive with or without Progesterone Receptors (PgR) positive, HER-negative) breast cancer who received adjuvant chemotherapy with positive lymph nodes or node-negative with tumor stage or pathological features according to Saint Gallen guidelines suggesting high-risk or when genomic testing determined in favor of adjuvant chemotherapy are eligible for registration in the study.

Before registration to the study, each patient signed an informed consent for the provision of biologic material for research purposes.

Potential biomarkers will be examined using in situ or molecular methods in Formalin fixed paraffin embedded (FFPE) tumor sections. For tumor subtyping immunohistochemistry for ER, PgR, HER2, Ki67 and Fluorescence in Situ Hybridization (FISH) will be performed where needed for the assessment of HER2 status; for Epidermal Growth Factor Receptor (EGFR) and CK5 for the classification of basal-like tumors; and, the expression of CD8, CD3 and FOXP3 on (Tumor- infiltrating Lymphocytes (TILs) will also be evaluated. Moreover, will be evaluated the mutational profile, including actionable genomic alterations, and the immune response -related profile of Greek women with breast cancer, via the application of DNA/RNA Next Generation Sequencing (NGS) technologies, relative also to patient outcome.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Luminal A breast cancer sub type
* Luminal B breast cancer sub type
* Positive lymph nodes
* Node- negative with tumor stage or pathological features according to Saint Gallen guidelines.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: This is a retrospective analysis of patients with operative early breast cancer of Luminal A and Luminal B sub types. Patients have been treated in Hellenic Cooperative Oncology Group (HeCOG) - affiliated departments of Oncology.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2013-04-24 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | From treatment initiation to the first documented disease progression, up to 5 years
Overall survival | From date of treatment initiation until death from any cause or date of last contact whichever occurred first, assessed up to 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: George Fountzilas, MD, Principal Investigator — Hellenic Cooperative Oncology Group
Locations (1):
- George Fountzilas, Athens, Greece

REFERENCES:
- [Background] Beguinot M, Dauplat MM, Kwiatkowski F, Lebouedec G, Tixier L, Pomel C, Penault-Llorca F, Radosevic-Robin N. Analysis of tumour-infiltrating lymphocytes reveals two new biologically different subgroups of breast ductal carcinoma in situ. BMC Cancer. 2018 Feb 3;18(1):129. doi: 10.1186/s12885-018-4013-6. PMID 29394917
- [Background] Burstein HJ, Curigliano G, Loibl S, Dubsky P, Gnant M, Poortmans P, Colleoni M, Denkert C, Piccart-Gebhart M, Regan M, Senn HJ, Winer EP, Thurlimann B; Members of the St. Gallen International Consensus Panel on the Primary Therapy of Early Breast Cancer 2019. Estimating the benefits of therapy for early-stage breast cancer: the St. Gallen International Consensus Guidelines for the primary therapy of early breast cancer 2019. Ann Oncol. 2019 Oct 1;30(10):1541-1557. doi: 10.1093/annonc/mdz235. PMID 31373601
- [Background] Ciriello G, Sinha R, Hoadley KA, Jacobsen AS, Reva B, Perou CM, Sander C, Schultz N. The molecular diversity of Luminal A breast tumors. Breast Cancer Res Treat. 2013 Oct;141(3):409-20. doi: 10.1007/s10549-013-2699-3. Epub 2013 Oct 6. PMID 24096568
- [Background] Curtis C, Shah SP, Chin SF, Turashvili G, Rueda OM, Dunning MJ, Speed D, Lynch AG, Samarajiwa S, Yuan Y, Graf S, Ha G, Haffari G, Bashashati A, Russell R, McKinney S; METABRIC Group; Langerod A, Green A, Provenzano E, Wishart G, Pinder S, Watson P, Markowetz F, Murphy L, Ellis I, Purushotham A, Borresen-Dale AL, Brenton JD, Tavare S, Caldas C, Aparicio S. The genomic and transcriptomic architecture of 2,000 breast tumours reveals novel subgroups. Nature. 2012 Apr 18;486(7403):346-52. doi: 10.1038/nature10983. PMID 22522925
- [Background] Diallo-Danebrock R, Ting E, Gluz O, Herr A, Mohrmann S, Geddert H, Rody A, Schaefer KL, Baldus SE, Hartmann A, Wild PJ, Burson M, Gabbert HE, Nitz U, Poremba C. Protein expression profiling in high-risk breast cancer patients treated with high-dose or conventional dose-dense chemotherapy. Clin Cancer Res. 2007 Jan 15;13(2 Pt 1):488-97. doi: 10.1158/1078-0432.CCR-06-1842. PMID 17255270
- [Background] Fountzilas G, Dafni U, Bobos M, Batistatou A, Kotoula V, Trihia H, Malamou-Mitsi V, Miliaras S, Chrisafi S, Papadopoulos S, Sotiropoulou M, Filippidis T, Gogas H, Koletsa T, Bafaloukos D, Televantou D, Kalogeras KT, Pectasides D, Skarlos DV, Koutras A, Dimopoulos MA. Differential response of immunohistochemically defined breast cancer subtypes to anthracycline-based adjuvant chemotherapy with or without paclitaxel. PLoS One. 2012;7(6):e37946. doi: 10.1371/journal.pone.0037946. Epub 2012 Jun 5. PMID 22679488
- [Background] Fountzilas G, Giannoulatou E, Alexopoulou Z, Zagouri F, Timotheadou E, Papadopoulou K, Lakis S, Bobos M, Poulios C, Sotiropoulou M, Lyberopoulou A, Gogas H, Pentheroudakis G, Pectasides D, Koutras A, Christodoulou C, Papandreou C, Samantas E, Papakostas P, Kosmidis P, Bafaloukos D, Karanikiotis C, Dimopoulos MA, Kotoula V. TP53 mutations and protein immunopositivity may predict for poor outcome but also for trastuzumab benefit in patients with early breast cancer treated in the adjuvant setting. Oncotarget. 2016 May 31;7(22):32731-53. doi: 10.18632/oncotarget.9022. PMID 27129168
- [Background] Gori S, Sidoni A, Colozza M, Ferri I, Mameli MG, Fenocchio D, Stocchi L, Foglietta J, Ludovini V, Minenza E, De Angelis V, Crino L. EGFR, pMAPK, pAkt and PTEN status by immunohistochemistry: correlation with clinical outcome in HER2-positive metastatic breast cancer patients treated with trastuzumab. Ann Oncol. 2009 Apr;20(4):648-54. doi: 10.1093/annonc/mdn681. Epub 2009 Feb 2. PMID 19188134
- [Background] Hammond ME, Hayes DF, Dowsett M, Allred DC, Hagerty KL, Badve S, Fitzgibbons PL, Francis G, Goldstein NS, Hayes M, Hicks DG, Lester S, Love R, Mangu PB, McShane L, Miller K, Osborne CK, Paik S, Perlmutter J, Rhodes A, Sasano H, Schwartz JN, Sweep FC, Taube S, Torlakovic EE, Valenstein P, Viale G, Visscher D, Wheeler T, Williams RB, Wittliff JL, Wolff AC; American Society of Clinical Oncology; College of American Pathologists. American Society of Clinical Oncology/College of American Pathologists guideline recommendations for immunohistochemical testing of estrogen and progesterone receptors in breast cancer (unabridged version). Arch Pathol Lab Med. 2010 Jul;134(7):e48-72. doi: 10.5858/134.7.e48. PMID 20586616
- [Background] Hendry S, Salgado R, Gevaert T, Russell PA, John T, Thapa B, Christie M, van de Vijver K, Estrada MV, Gonzalez-Ericsson PI, Sanders M, Solomon B, Solinas C, Van den Eynden GGGM, Allory Y, Preusser M, Hainfellner J, Pruneri G, Vingiani A, Demaria S, Symmans F, Nuciforo P, Comerma L, Thompson EA, Lakhani S, Kim SR, Schnitt S, Colpaert C, Sotiriou C, Scherer SJ, Ignatiadis M, Badve S, Pierce RH, Viale G, Sirtaine N, Penault-Llorca F, Sugie T, Fineberg S, Paik S, Srinivasan A, Richardson A, Wang Y, Chmielik E, Brock J, Johnson DB, Balko J, Wienert S, Bossuyt V, Michiels S, Ternes N, Burchardi N, Luen SJ, Savas P, Klauschen F, Watson PH, Nelson BH, Criscitiello C, O'Toole S, Larsimont D, de Wind R, Curigliano G, Andre F, Lacroix-Triki M, van de Vijver M, Rojo F, Floris G, Bedri S, Sparano J, Rimm D, Nielsen T, Kos Z, Hewitt S, Singh B, Farshid G, Loibl S, Allison KH, Tung N, Adams S, Willard-Gallo K, Horlings HM, Gandhi L, Moreira A, Hirsch F, Dieci MV, Urbanowicz M, Brcic I, Korski K, Gaire F, Koeppen H, Lo A, Giltnane J, Rebelatto MC, Steele KE, Zha J, Emancipator K, Juco JW, Denkert C, Reis-Filho J, Loi S, Fox SB. Assessing Tumor-infiltrating Lymphocytes in Solid Tumors: A Practical Review for Pathologists and Proposal for a Standardized Method From the International Immunooncology Biomarkers Working Group: Part 1: Assessing the Host Immune Response, TILs in Invasive Breast Carcinoma and Ductal Carcinoma In Situ, Metastatic Tumor Deposits and Areas for Further Research. Adv Anat Pathol. 2017 Sep;24(5):235-251. doi: 10.1097/PAP.0000000000000162. PMID 28777142
- [Background] Kennecke H, Yerushalmi R, Woods R, Cheang MC, Voduc D, Speers CH, Nielsen TO, Gelmon K. Metastatic behavior of breast cancer subtypes. J Clin Oncol. 2010 Jul 10;28(20):3271-7. doi: 10.1200/JCO.2009.25.9820. Epub 2010 May 24. PMID 20498394
- [Background] Kim JY, Lee E, Park K, Park WY, Jung HH, Ahn JS, Im YH, Park YH. Immune signature of metastatic breast cancer: Identifying predictive markers of immunotherapy response. Oncotarget. 2017 Jul 18;8(29):47400-47411. doi: 10.18632/oncotarget.17653. PMID 28537889
- [Background] Koletsa T, Kotoula V, Koliou GA, Manousou K, Chrisafi S, Zagouri F, Sotiropoulou M, Pentheroudakis G, Papoudou-Bai A, Christodoulou C, Xepapadakis G, Zografos G, Petraki K, Pazarli E, Koutras A, Kourea HP, Bafaloukos D, Chatzopoulos K, Iliadis A, Markopoulos C, Venizelos V, Arnogiannaki N, Kalogeras KT, Kostopoulos I, Gogas H, Fountzilas G. Prognostic impact of stromal and intratumoral CD3, CD8 and FOXP3 in adjuvantly treated breast cancer: do they add information over stromal tumor-infiltrating lymphocyte density? Cancer Immunol Immunother. 2020 Aug;69(8):1549-1564. doi: 10.1007/s00262-020-02557-0. Epub 2020 Apr 18. PMID 32303794
- [Background] Lim E, Winer EP. Adjuvant chemotherapy in luminal breast cancers. Breast. 2011 Oct;20 Suppl 3:S128-31. doi: 10.1016/S0960-9776(11)70309-5. PMID 22015279
- [Background] Cancer Genome Atlas Network. Comprehensive molecular portraits of human breast tumours. Nature. 2012 Oct 4;490(7418):61-70. doi: 10.1038/nature11412. Epub 2012 Sep 23. PMID 23000897
- [Background] Paluch BE, Glenn ST, Conroy JM, Papanicolau-Sengos A, Bshara W, Omilian AR, Brese E, Nesline M, Burgher B, Andreas J, Odunsi K, Eng K, He J, Qin M, Gardner M, Galluzzi L, Morrison CD. Robust detection of immune transcripts in FFPE samples using targeted RNA sequencing. Oncotarget. 2017 Jan 10;8(2):3197-3205. doi: 10.18632/oncotarget.13691. PMID 27911273
- [Background] Prat A, Perou CM. Deconstructing the molecular portraits of breast cancer. Mol Oncol. 2011 Feb;5(1):5-23. doi: 10.1016/j.molonc.2010.11.003. Epub 2010 Nov 24. PMID 21147047
- [Background] Press MF, Sauter G, Buyse M, Bernstein L, Guzman R, Santiago A, Villalobos IE, Eiermann W, Pienkowski T, Martin M, Robert N, Crown J, Bee V, Taupin H, Flom KJ, Tabah-Fisch I, Pauletti G, Lindsay MA, Riva A, Slamon DJ. Alteration of topoisomerase II-alpha gene in human breast cancer: association with responsiveness to anthracycline-based chemotherapy. J Clin Oncol. 2011 Mar 1;29(7):859-67. doi: 10.1200/JCO.2009.27.5644. Epub 2010 Dec 28. PMID 21189395
- [Background] Romero Q, Bendahl PO, Ferno M, Grabau D, Borgquist S. A novel model for Ki67 assessment in breast cancer. Diagn Pathol. 2014 Jun 16;9:118. doi: 10.1186/1746-1596-9-118. PMID 24934660
- [Background] Rouzier R, Perou CM, Symmans WF, Ibrahim N, Cristofanilli M, Anderson K, Hess KR, Stec J, Ayers M, Wagner P, Morandi P, Fan C, Rabiul I, Ross JS, Hortobagyi GN, Pusztai L. Breast cancer molecular subtypes respond differently to preoperative chemotherapy. Clin Cancer Res. 2005 Aug 15;11(16):5678-85. doi: 10.1158/1078-0432.CCR-04-2421. PMID 16115903
- [Background] Safonov A, Jiang T, Bianchini G, Gyorffy B, Karn T, Hatzis C, Pusztai L. Immune Gene Expression Is Associated with Genomic Aberrations in Breast Cancer. Cancer Res. 2017 Jun 15;77(12):3317-3324. doi: 10.1158/0008-5472.CAN-16-3478. Epub 2017 Apr 20. PMID 28428277
- [Background] Shah SP, Roth A, Goya R, Oloumi A, Ha G, Zhao Y, Turashvili G, Ding J, Tse K, Haffari G, Bashashati A, Prentice LM, Khattra J, Burleigh A, Yap D, Bernard V, McPherson A, Shumansky K, Crisan A, Giuliany R, Heravi-Moussavi A, Rosner J, Lai D, Birol I, Varhol R, Tam A, Dhalla N, Zeng T, Ma K, Chan SK, Griffith M, Moradian A, Cheng SW, Morin GB, Watson P, Gelmon K, Chia S, Chin SF, Curtis C, Rueda OM, Pharoah PD, Damaraju S, Mackey J, Hoon K, Harkins T, Tadigotla V, Sigaroudinia M, Gascard P, Tlsty T, Costello JF, Meyer IM, Eaves CJ, Wasserman WW, Jones S, Huntsman D, Hirst M, Caldas C, Marra MA, Aparicio S. The clonal and mutational evolution spectrum of primary triple-negative breast cancers. Nature. 2012 Apr 4;486(7403):395-9. doi: 10.1038/nature10933. PMID 22495314
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2020. CA Cancer J Clin. 2020 Jan;70(1):7-30. doi: 10.3322/caac.21590. Epub 2020 Jan 8. PMID 31912902
- [Background] Smid M, Rodriguez-Gonzalez FG, Sieuwerts AM, Salgado R, Prager-Van der Smissen WJ, Vlugt-Daane MV, van Galen A, Nik-Zainal S, Staaf J, Brinkman AB, van de Vijver MJ, Richardson AL, Fatima A, Berentsen K, Butler A, Martin S, Davies HR, Debets R, Gelder ME, van Deurzen CH, MacGrogan G, Van den Eynden GG, Purdie C, Thompson AM, Caldas C, Span PN, Simpson PT, Lakhani SR, Van Laere S, Desmedt C, Ringner M, Tommasi S, Eyford J, Broeks A, Vincent-Salomon A, Futreal PA, Knappskog S, King T, Thomas G, Viari A, Langerod A, Borresen-Dale AL, Birney E, Stunnenberg HG, Stratton M, Foekens JA, Martens JW. Breast cancer genome and transcriptome integration implicates specific mutational signatures with immune cell infiltration. Nat Commun. 2016 Sep 26;7:12910. doi: 10.1038/ncomms12910. PMID 27666519
- [Background] Sorlie T, Perou CM, Tibshirani R, Aas T, Geisler S, Johnsen H, Hastie T, Eisen MB, van de Rijn M, Jeffrey SS, Thorsen T, Quist H, Matese JC, Brown PO, Botstein D, Lonning PE, Borresen-Dale AL. Gene expression patterns of breast carcinomas distinguish tumor subclasses with clinical implications. Proc Natl Acad Sci U S A. 2001 Sep 11;98(19):10869-74. doi: 10.1073/pnas.191367098. PMID 11553815
- [Background] Stephens PJ, Tarpey PS, Davies H, Van Loo P, Greenman C, Wedge DC, Nik-Zainal S, Martin S, Varela I, Bignell GR, Yates LR, Papaemmanuil E, Beare D, Butler A, Cheverton A, Gamble J, Hinton J, Jia M, Jayakumar A, Jones D, Latimer C, Lau KW, McLaren S, McBride DJ, Menzies A, Mudie L, Raine K, Rad R, Chapman MS, Teague J, Easton D, Langerod A; Oslo Breast Cancer Consortium (OSBREAC); Lee MT, Shen CY, Tee BT, Huimin BW, Broeks A, Vargas AC, Turashvili G, Martens J, Fatima A, Miron P, Chin SF, Thomas G, Boyault S, Mariani O, Lakhani SR, van de Vijver M, van 't Veer L, Foekens J, Desmedt C, Sotiriou C, Tutt A, Caldas C, Reis-Filho JS, Aparicio SA, Salomon AV, Borresen-Dale AL, Richardson AL, Campbell PJ, Futreal PA, Stratton MR. The landscape of cancer genes and mutational processes in breast cancer. Nature. 2012 May 16;486(7403):400-4. doi: 10.1038/nature11017. PMID 22722201
- [Background] Vanden Bempt I, Van Loo P, Drijkoningen M, Neven P, Smeets A, Christiaens MR, Paridaens R, De Wolf-Peeters C. Polysomy 17 in breast cancer: clinicopathologic significance and impact on HER-2 testing. J Clin Oncol. 2008 Oct 20;26(30):4869-74. doi: 10.1200/JCO.2007.13.4296. Epub 2008 Sep 15. PMID 18794552
- [Background] Wolff AC, Hammond ME, Schwartz JN, Hagerty KL, Allred DC, Cote RJ, Dowsett M, Fitzgibbons PL, Hanna WM, Langer A, McShane LM, Paik S, Pegram MD, Perez EA, Press MF, Rhodes A, Sturgeon C, Taube SE, Tubbs R, Vance GH, van de Vijver M, Wheeler TM, Hayes DF; American Society of Clinical Oncology; College of American Pathologists. American Society of Clinical Oncology/College of American Pathologists guideline recommendations for human epidermal growth factor receptor 2 testing in breast cancer. J Clin Oncol. 2007 Jan 1;25(1):118-45. doi: 10.1200/JCO.2006.09.2775. Epub 2006 Dec 11. PMID 17159189